CLINICAL TRIAL: NCT00562185
Title: A Phase I/II Study of Intravenous Doxil and Intraperitoneal Carboplatin as Salvage Therapy in Patients With Recurrent Ovarian Cancer
Brief Title: Doxorubicin and Carboplatin in Treating Patients With Recurrent Ovarian Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding source withdrew funding
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Ortho Biotech Clinical Affairs, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000574034; SCCC-04E07; SCCC-062007-043; ORTHO-SCCC-04E07
Record Dates: First submitted 2007-11-20; First posted 2007-11-21 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-10

CONDITIONS: Ovarian Cancer
Keywords: recurrent ovarian epithelial cancer; ovarian sarcoma; recurrent ovarian germ cell tumor; ovarian stromal cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Carboplatin; Doxorubicin

INTERVENTIONS:
Drug: carboplatin
Drug: doxorubicin hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as doxorubicin and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving doxorubicin together with carboplatin may kill more tumor cells.

PURPOSE: This phase I and phase II trial is studying the side effects and best dose of carboplatin when given together with doxorubicin to see how well it works in treating patients with recurrent ovarian cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum tolerated dose and safety of intravenous doxorubicin hydrochloride and intraperitoneal carboplatin in patients with platinum-sensitive recurrent ovarian cancer.
* To evaluate the feasibility of this regimen in these patients.

Secondary

* To evaluate the response rate and progression-free survival of patients with recurrent ovarian cancer who have had no more than two prior salvage regimens.

OUTLINE: This is a phase I dose-escalation study of carboplatin followed by a phase II study.

* Phase I: Patients receive doxorubicin hydrochloride IV over 1 hour followed by carboplatin intraperitoneally on day 1 until the maximum tolerated dose is achieved. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
* Phase II: Patients receive doxorubicin hydrochloride as in phase I and carboplatin at the maximum tolerated dose as in phase I.

After completion of study treatment, patients are followed every 4 weeks for 1 year.

PROJECTED ACCRUAL: A total of 61 patients (18 patients in phase I and 43 patients in phase II) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ovarian carcinoma

  * Recurrent disease
* Known platinum-sensitive recurrent disease after no more than 2 prior salvage regimens
* Measurable disease as defined by a target lesion and a CA125 level
* No epithelial ovarian carcinoma of low malignant potential

PATIENT CHARACTERISTICS:

Inclusion criteria:

* GOG performance status 0, 1, or 2
* Life expectancy > 6 months
* Absolute neutrophil count ≥ 1,500/uL
* Platelet count ≥ 100,000/uL
* Hemoglobin > 9.0 g/dL
* Creatinine ≤ 2.0 mg/dL
* Bilirubin ≤ 1.5 x upper limit of normal (ULN)
* SGOT and alkaline phosphatase ≤ 3 x ULN
* Neuropathy (sensory and motor) ≤ CTCAE grade 1

Exclusion criteria:

* GOG performance status 3 or 4
* Pregnant or breastfeeding
* History of hypersensitivity reactions attributed to a conventional formulation of doxorubicin hydrochloride or the components of DOXIL®
* Abnormal LVEF as determined by gated cardiac radionucleotide scan (MUGA)
* Septicemia or severe infection
* Acute hepatitis or severe gastrointestinal bleeding
* Any of the following:

  * Unstable angina
  * Myocardial infarction within the past 6 months
  * NYHA class II-IV heart failure
  * Uncontrolled angina
  * Severe uncontrolled ventricular arrhythmias
  * Clinically significant pericardial disease
  * Electrocardiographic evidence of acute ischemic or active conduction system abnormalities

    * Patients with evidence of abnormal cardiac conduction (e.g., bundle branch block or heart block) are eligible if their disease has been stable for the past six months
* Other invasive malignancies within the past 5 years except for nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

Inclusion criteria:

* See Disease Characteristics
* At least 6 months since prior adjuvant regimen
* At least 4 weeks since prior salvage treatment
* May have received secondary cytoreduction for recurrent ovarian cancer
* May have received prior intraperitoneal therapy for ovarian cancer
* May have received no more than 2 prior platinum and taxane-based regimens
* May have received prior intraperitoneal platinum during front-line treatment

Exclusion criteria:

* Prior anthracycline dose exceeding 360 mg/m^2 for doxorubicin hydrochloride (including DOXIL®) or 720 mg/m^2 for epirubicin hydrochloride
* Prior radiotherapy
* Prior intraperitoneal carboplatin or cisplatin as salvage treatment for recurrent ovarian cancer
* Concurrent amifostine or other protective agents

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Acute toxicity
Maximum tolerated dose of intraperitoneal carboplatin when given in combination with IV doxorubicin hydrochloride (phase I)
Primary efficacy and safety (phase II)

CONTACTS AND LOCATIONS:
Overall Officials: Jayanthi S. Lea, MD, Study Chair — Simmons Cancer Center
Locations (1):
- Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas, United States